CLINICAL TRIAL: NCT02801201
Title: Impact of Analgesia on Success of External Version: Comparison of Spinal Anesthesia Versus Sedation; Prospective, Controlled, Randomized Study
Brief Title: Impact of Analgesia on Success of External Version: Comparison of Spinal Anesthesia Versus Sedation
Acronym: RaVem
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2016_843_0001
Record Dates: First submitted 2016-05-27; First posted 2016-06-15 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Breech Presentation
Keywords: sedation; spinal anesthesia
MeSH Terms: conditions — Breech Presentation | interventions — Midazolam; Bupivacaine

ARMS (2):
- sedation (Active Comparator): Midazolam : 0,10 mg/kg
  Interventions: Drug: Midazolam
- spinal anesthesia (Active Comparator): Bupivacain 10 mg
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Midazolam
  Arms: sedation
Drug: Bupivacaine
  Arms: spinal anesthesia

SUMMARY:
At the time of birth, nearly 5% of children are in breech presentation. This type of presentation requires a medical environment and leads to more frequent use of Caesarean sections. This is why the external version can be proposed, usually from the 36th week. Its success rate is 40%, and is usually performed under simple sedation. One of the causes of failure is the lack of relaxation of the uterus, which could be higher in case of deeper anesthesia, as is the case in spinal anesthesia. The study project is to demonstrate superiority of spinal anesthesia compared to the usual protocol sedation in terms of primary and secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* patient with 36 weeks of amenorrhea (SA) a fetus breech or transverse presentation
* covered by a an insurance system
* signed contentment

Exclusion Criteria:

Obstetric contraindications:

* placenta previa
* 3rd trimester bleeding
* suspicion of fetal anoxia
* patient has already received more than one caesarean section
* multi-fetal pregnancy
* HIV +
* anticoagulant therapy

Anesthesiologic contraindications:

* infection at the puncture site, systemic infection or severe sepsis
* intracranial hypertension
* uncompensated heart failure
* constitute or acquired coagulation abnormalities, including anticoagulant therapy with curative intent
* neuropathy with demyelination of nerve fibers in thrust or unstabilized during recovery
* syringomyelia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-05-31 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Successful external version (VME) upon completion gesture : obtaining a fetus in cephalic presentation | 24 hours

SECONDARY OUTCOMES:
occurrence of side events due to the manipulation itself | Day 0
  cesarean for non resolutive bradycardia, placental abruption, rupture of amniotic membranes
occurrence of side events due to anesthesia | Day 0
  hypotension, maternal bradycardia, desaturation, nausea / vomiting, number of punctures greater than 1 (failure of the first puncture for spinal anesthesia leading to the necessity to perform one or more others).
The pain experienced by the patient: assessed by the Visual Analogic Scale | Day 0
The final delivery mode (caesarian section or vaginal) | Day 0
The presentation in childbirth | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Julien CHEVREAU, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France